CLINICAL TRIAL: NCT01435135
Title: Randomized, Double Blind Evaluation of Late Boost Strategies for HIV-uninfected Participants in the HIV Vaccine Efficacy Trial RV 144: "Aventis Pasteur Live Recombinant ALVAC-HIV (vCP1521) Priming With VaxGen gp120 B/E (AIDSVAX B/E) Boosting in HIV-uninfected Thai Adults"
Brief Title: Study of Late Boost Strategies for HIV-uninfected Participants From Protocol RV 144
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RV 305; WRAIR #1792 (Other: WRAIR IRB); A-14430.13 (Other: USAMRMC HRPO); S-10-0010 (Other: Sponsor)
Record Dates: First submitted 2011-09-08; First posted 2011-09-15 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — AIDSVAX; AIDSVAX B-E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group I (Experimental): ALVAC-HIV + AIDSVAX B/E or ALVAC-HIV placebo + AIDSVAX B/E placebo at Weeks 0 and 24
  Interventions: Biological: ALVAC-HIV; Biological: AIDSVAX B/E; Biological: ALVAC-HIV Placebo; Biological: AIDSVAX B/E Placebo
- Group II (Experimental): AIDSVAX B/E or AIDSVAX B/E placebo at Weeks 0 and 24
  Interventions: Biological: AIDSVAX B/E; Biological: AIDSVAX B/E Placebo
- Group III (Experimental): ALVAC-HIV or ALVAC-HIV placebo at Weeks 0 and 24
  Interventions: Biological: ALVAC-HIV; Biological: ALVAC-HIV Placebo

INTERVENTIONS:
Biological: ALVAC-HIV — 1 mL per injection containing 10^6 CCID50/dose administered
  Other Names: (vCP1521)
  Arms: Group I; Group III
Biological: AIDSVAX B/E — 1 mL per injection (300 ug dose/antigen for a total of 600ug/dose administered)
  Arms: Group I; Group II
Biological: ALVAC-HIV Placebo — 1 ml per injection
  Arms: Group I; Group III
Biological: AIDSVAX B/E Placebo — 1 ml per injection
  Arms: Group I; Group II

SUMMARY:
The purpose of this study is to assess safety and tolerability of late boost regimens of AIDSVAX B/E alone, ALVAC-HIV alone, or ALVAC-HIV/AIDSVAX B/E combination in HIV-uninfected participants from RV 144.

ELIGIBILITY:
Inclusion Criteria:

* Must have participated in RV144, received the active product, and completed all 4 vaccination visits per protocol.
* Must be able to understand and complete the informed consent process.
* Must successfully complete a Test of Understanding prior to enrollment

  * The volunteer must answer 80% or 8 out of 10 of the questions correctly including two compulsory questions answered correctly.
  * If the volunteer is unable to do so, he or she will be given two more opportunities to repeat the TOU.
  * If after three attempts to pass the TOU the volunteer is still unable to do so, the volunteer will become ineligible for study participation.
* Must be in good general health without clinically significant medical history.
* HIV-uninfected per predefined algorithm within 45 days of enrollment.
* Laboratory screening analysis

  * Hemoglobin: Women ≥12.0 g/dL. Men ≥12.5 g/dL
  * White cell count: 4,000 to 11,000 cells/mm3
  * Platelets: 150,000 to 450,000/mm3
  * Normal liver function: ALT/AST ≤1.25 institutional upper limit of reference range
  * Creatinine: ≤1.25 institutional upper limit of reference range
* Urinalysis (dipstick) for blood and protein no greater than 1+, glucose negative
* Female-Specific Criteria:

  * Negative human choriogonadotropin (β-HCG) pregnancy test (urine) for women prior to each vaccination (same day).
  * Be using adequate birth control methods for 45 days prior to the first vaccine/placebo vaccination and will continue to be followed for at least 3 months after the final vaccine/placebo vaccination. Adequate birth control is defined as follows: Contraceptive medications delivered orally, intramuscularly, vaginally, or implanted underneath the skin, surgical methods (hysterectomy or bilateral tubal ligation), condoms, diaphragms, intrauterine device (IUD), abstinence.

Exclusion Criteria:

1. Women breast-feeding or pregnant (positive pregnancy test) or planning to become pregnant during the window between study enrollment and 3 months after the last vaccination visit.

* History of anaphylaxis or other serious adverse reaction to vaccines including to RV 144 vaccines, or allergies or reactions likely to be exacerbated by any component of the vaccine or placebo, including eggs, egg products, streptomycin, or neomycin.
* Subject has received any of the following substances:

  * Chronic use of therapies which may modify immune response, such as IV immune globulin and systemic corticosteroids (in doses of > 20 mg/day prednisone equivalent for periods exceeding 10 days).
  * The following exceptions are permitted and will not exclude study participation: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis; or a short course (duration of 10 days or less, or a single injection) of corticosteroid for a nonchronic condition (based on investigator clinical judgment) at least 2 weeks prior to enrollment in this study.
  * Blood products within 120 days prior to HIV screening.
  * Immunoglobulins within 14 days prior to HIV screening.
  * Any vaccine within 14 days prior to initial study vaccine administration in the present study.
  * Receipt of investigational HIV vaccine product other than the RV 144 regimen.
  * Investigational research agents within 30 days prior to initial study vaccine administration in the present study.
  * Use of anti-tuberculosis prophylaxis or therapy during the past 90 days.
* Any medical, psychiatric, social condition, occupational reason, or other responsibility that, in the judgment of the investigator, is a contraindication to protocol compliance or impairs a subject's ability to give informed consent.
* Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within 5 years prior to enrollment, a history of suicide plan or attempt.
* Study site employees who are involved in the protocol and/or may have direct access to study related area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2012-04 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Primary Immunogenicity Endpoint | Week 0
  Characterization of vaccine-induced immune responses by IFN-gamma ELISPOT, intracellular cytokine staining (ICS), and 3H-thymidine incorporation assay.
Safety Endpoints | During the 3 days post-vaccination
  Post-vaccination reactions including erythema, induration, pain/tenderness, swelling, limitation of arm movement, fever, tiredness, chills, myalgia, arthralgia, headache, nausea, dizziness, and rash will be assessed and recorded on diary cards.
Primary Immunogenicity Endpoint | Week 2
  Characterization of vaccine-induced immune responses by IFN-gamma ELISPOT, intracellular cytokine staining (ICS), and 3H-thymidine incorporation assay.
Primary Immunogenicity Endpoint | Week 24
  Characterization of vaccine-induced immune responses by IFN-gamma ELISPOT, intracellular cytokine staining (ICS), and 3H-thymidine incorporation assay.
Primary Immunogenicity Endpoint | Week 26
  Characterization of vaccine-induced immune responses by IFN-gamma ELISPOT, intracellular cytokine staining (ICS), and 3H-thymidine incorporation assay.
Primary Immunogenicity Endpoint | Week 48
  Characterization of vaccine-induced immune responses by IFN-gamma ELISPOT, intracellular cytokine staining (ICS), and 3H-thymidine incorporation assay.
Primary Immunogenicity Endpoint | Week 72
  Characterization of vaccine-induced immune responses by IFN-gamma ELISPOT, intracellular cytokine staining (ICS), and 3H-thymidine incorporation assay.

SECONDARY OUTCOMES:
Secondary Immunogenicity Endpoints | Baseline, Weeks 2, 24, 26, 48 and 72
  Characterization of vaccine-induced immune responses by lymphoproliferation assays (LPA), human leukocyte antigen (HLA) subtyping, characterization of natural killer (NK) cells using multiparameter flow, assessment of APOBEC 3G (A3G) antiretroviral factor expression, B-cell ELISPOT, HIV-specific binding antibody assays, neutralizing antibody assays, mucosal IgG and IgA binding antibody assays, antibody-dependent cell mediated cytotoxicity (ADCC) and antibody-dependent cell mediated viral inhibition (ADCVI) assays

CONTACTS AND LOCATIONS:
Overall Officials: Supachai Rerks-Ngarm, MD, Principal Investigator — Department of Disease Control, Ministry of Public Health, Nonthaburi, Thailand
Locations (2):
- Thailand (2):
  - Bang Lamung District Hospital, Chon Buri
  - Phan Thong District Hospital, Chon Buri

REFERENCES:
- [Background] Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Kaewkungwal J, Chiu J, Paris R, Premsri N, Namwat C, de Souza M, Adams E, Benenson M, Gurunathan S, Tartaglia J, McNeil JG, Francis DP, Stablein D, Birx DL, Chunsuttiwat S, Khamboonruang C, Thongcharoen P, Robb ML, Michael NL, Kunasol P, Kim JH; MOPH-TAVEG Investigators. Vaccination with ALVAC and AIDSVAX to prevent HIV-1 infection in Thailand. N Engl J Med. 2009 Dec 3;361(23):2209-20. doi: 10.1056/NEJMoa0908492. Epub 2009 Oct 20. PMID 19843557
- [Derived] Williams LD, Shen X, Sawant SS, Akapirat S, Dahora LC, Tay MZ, Stanfield-Oakley S, Wills S, Goodman D, Tenney D, Spreng RL, Zhang L, Yates NL, Montefiori DC, Eller MA, Easterhoff D, Hope TJ, Rerks-Ngarm S, Pittisuttithum P, Nitayaphan S, Excler JL, Kim JH, Michael NL, Robb ML, O'Connell RJ, Karasavvas N, Vasan S, Ferrari G, Tomaras GD; RV305 study team. Viral vector delivered immunogen focuses HIV-1 antibody specificity and increases durability of the circulating antibody recall response. PLoS Pathog. 2023 May 31;19(5):e1011359. doi: 10.1371/journal.ppat.1011359. eCollection 2023 May. PMID 37256916
- [Derived] Rerks-Ngarm S, Pitisuttithum P, Excler JL, Nitayaphan S, Kaewkungwal J, Premsri N, Kunasol P, Karasavvas N, Schuetz A, Ngauy V, Sinangil F, Dawson P, deCamp AC, Phogat S, Garunathan S, Tartaglia J, DiazGranados C, Ratto-Kim S, Pegu P, Eller M, Karnasuta C, Montefiori DC, Sawant S, Vandergrift N, Wills S, Tomaras GD, Robb ML, Michael NL, Kim JH, Vasan S, O'Connell RJ; RV305 Study Team. Randomized, Double-Blind Evaluation of Late Boost Strategies for HIV-Uninfected Vaccine Recipients in the RV144 HIV Vaccine Efficacy Trial. J Infect Dis. 2017 Apr 15;215(8):1255-1263. doi: 10.1093/infdis/jix099. PMID 28329190
- [Derived] Easterhoff D, Moody MA, Fera D, Cheng H, Ackerman M, Wiehe K, Saunders KO, Pollara J, Vandergrift N, Parks R, Kim J, Michael NL, O'Connell RJ, Excler JL, Robb ML, Vasan S, Rerks-Ngarm S, Kaewkungwal J, Pitisuttithum P, Nitayaphan S, Sinangil F, Tartaglia J, Phogat S, Kepler TB, Alam SM, Liao HX, Ferrari G, Seaman MS, Montefiori DC, Tomaras GD, Harrison SC, Haynes BF. Boosting of HIV envelope CD4 binding site antibodies with long variable heavy third complementarity determining region in the randomized double blind RV305 HIV-1 vaccine trial. PLoS Pathog. 2017 Feb 24;13(2):e1006182. doi: 10.1371/journal.ppat.1006182. eCollection 2017 Feb. PMID 28235027